CLINICAL TRIAL: NCT06660212
Title: Is Multimodal Physiotherapy And/or Photobiomodulation Therapy Effective for Pain Reduction Among Those Who Experience Provoked Vestibulodynia: a Randomized Controlled Trial
Brief Title: Biomodulation and Rehabilitation Interventions to TarGet Pelvic Health
Acronym: BRIGHT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); University of Laval, Quebec City, Canada (Unknown); BioFlexTM Laser Therapy (Unknown)
Responsible Party: Principal Investigator, Dr. Linda McLean, Professor, University of Ottawa
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-08-24-10662
Record Dates: First submitted 2024-10-23; First posted 2024-10-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-10

CONDITIONS: Vulvodynia; Provoked Vestibulodynia; Dyspareunia
Keywords: Provoked vestibulodynia; Intervention; Vulvodynia; Double-blinded; Pelvic floor; laser; Vulvar pain
MeSH Terms: conditions — Vulvodynia; Dyspareunia | interventions — Low-Level Light Therapy; Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: 2x2 factorial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants and investigators in this 2x2 factorial clinical trial will be blinded through a process of random allocation managed by a third-party investigator who is not involved in the direct administration of treatments or outcome assessments. This third-party investigator will use a computerized randomization system to assign participants to one of the four treatment groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Sham laser (Sham Comparator): 15 treatments will be provided over a 14 week period but at an intensity of 1% output for all sites and at all stages. Each treatment will last approximately 20 minutes. At each visit, the array will be applied to the surface of the perineum (red and infrared light), followed by treatment at specific painful sites using the red light probe.
  Interventions: Device: Sham photobiomodulation
- Real laser (Active Comparator): 15 treatments will be provided over a 14 week period. Each treatment will last approximately 20 minutes and will include the laser array first being applied to the surface of the perineum (red and infrared light) and the focal probe will be applied to painful sites on the perineum. All the stages will involve use of the same array and probe placement, but at each stage the dosage will be increased according to the BioFlex protocol.
  Interventions: Device: Photobiomodulation
- Sham laser + multi-modal physiotherapy (Active Comparator): Over 14 weeks, participants will receive 10 physiotherapy sessions and 15 sham laser sessions, lasting a total of 50 minutes. Laser and physiotherapy treatments will be delivered within the same visit where possible. For the physiotherapy, the therapist will start with education, followed by progressive relaxation exercises and deep breathing. Participants will practice graded pelvic floor muscle (PFM) contractions, manual stretching techniques with external palpation, and gradually progressing to the insertion of one or two fingers into the vagina. Finally, vaginal dilators will be used to stretch the vaginal opening and PFMs. The participant will use relaxation breathing and contraction/relaxation cycles to facilitate insertion, progressing to larger dilators as tolerated. For the sham laser, the same protocol will be followed as described in previous arms.
  Interventions: Device: Sham photobiomodulation; Procedure: Multimodal physiotherapy
- Laser + multi-modal physiotherapy (Experimental): This treatment group will receive a combination therapy (i.e., both laser and physiotherapy), with each session lasting up to 50 minutes over a 14 week period. Laser and physiotherapy treatments will be delivered within the same visit where possible. Laser and physiotherapy protocols will be delivered as described in the previous arms.
  Interventions: Device: Photobiomodulation; Procedure: Multimodal physiotherapy

INTERVENTIONS:
Device: Photobiomodulation — The laser therapy will be delivered in progressively higher doses, based on individual participants. Each stage will follow this sequence of applications: (1) perineum application (DUO-240 red and infrared array in the surface of the perineum) and (2) LDR-100 probe on the vestibula more generally. Doses will increase from 40%-100% power over the course of the intervention
  Other Names: Low level laser therapy
  Arms: Laser + multi-modal physiotherapy; Real laser
Device: Sham photobiomodulation — The laser therapy will be delivered in progressively higher doses, based on individual participants tolerance. Each stage will follow this sequence of applications: (1) perineum application (DUO-240 red and infrared array in the surface of the perineum) and (2) LDR-100 probe on the vestibula more generally. . Doses will always be set to 1% power over the course of the intervention
  Arms: Sham laser; Sham laser + multi-modal physiotherapy
Procedure: Multimodal physiotherapy — A total of 10 sessions of multimodal physiotherapy interventions will be provided to each of the participants in the multimodal physiotherapy (mPT) and multimodal physiotherapy combined with photobiomodulation treatment (mPT+PBM) groups. In general, each session will take place in the following order:1) Subjective assessment of the condition and screening for adverse effects or deterioration of the condition, 2)Education, 3) Relaxation Techniques, 4) Pelvic Floor Muscle Exercises, 5) Manual techniques, 6) exercises with accommodators, 7) Global exercises, 8) Assessment of the post-treatment condition and 9) adjustment of the weekly exercise program to be done at home. Each of these 9 treatments will be adjusted and tailored to each participant and progressed based on individual preference and response to treatment under the discretion of the study physiotherapist.
  Other Names: Physiotherapy
  Arms: Laser + multi-modal physiotherapy; Sham laser + multi-modal physiotherapy

SUMMARY:
This trial will provide evidence for the effective management of pain and pain-related domains among those who experience provoked vestibulodynia (PVD) using photobiomodulation (PBM) and multimodal physiotherapy (mPT) in a randomized controlled trial (RCT). PVD is the most common subcategory of vulvovaginal pain experienced during sexual and non-sexual activities, affects the psychological and sexual health of an astounding one in five Canadian women, yet access to evidence-informed management approaches is limited. We will employ four intervention groups: PBM, sham PBM (control), PBM combined with mPT, and mPT with sham PBM to evaluate the effectiveness of each approach on its own and the two approaches in combination.

Among those who experience PVD, we seek to answer:

1. Relative to baseline and to sham PBM, does a 14-week intervention involving PBM, mPT, or a combination of mPT and PMB reduce vulvar pain severity reported on the Vulvar Pain Assessment Questionnaire (VPAQ)?
2. Is a combined mPT and PBM intervention more effective than mPT or PMB alone when considering vulvar pain severity and/or related domains as measured through VPAQ?
3. Are positive changes in vulvar pain severity and related domains observed following a 14-week intervention involving PBM, mPT or a combination of PBM and mPT retained at 6 months and at 1 year?

Secondary objectives include determining the effectiveness of PBM, mPT, and mPT combined with PBM relative to sham PBM on: Patient Global Impression of Change (PGIC), pain sensitivity measured using provocative tests, the other domains of the VPAQ, sexual function, as well as investigating mediating effects of psychosocial variables (central sensitization index, chronic pain acceptance), gender identity, and the presence of vaginismus on patient response to mPT, PBM and mPT combined with PBM. Lastly we will monitor patient satisfaction with the interventions, adherence to the interventions, and any adverse events.

DETAILED DESCRIPTION:
Despite its high prevalence, surprisingly little is known about vulvovaginal pain in general and PVD more specifically. It is characterized by severe sharp and/or burning pain at the entrance to the vagina (i.e. the vulvar vestibule) when pressure is applied to it and it has been primarily attributed to inflammatory processes, hyper-innervation, and pelvic floor muscle (PFM) overactivity.

While it remains under-reported due to embarrassment and shame, the prevalence of PVD in premenopausal women is estimated at 12%, who account for 87% of cases. PVD pain can be intense and can last for days following attempts at sexual and non-sexual (e.g., tampon insertion) activities. It negatively impacts the physical, social and sexual health of women who experience it, and it can have major implications for reproductive health including functional infertility when those affected are unable to have penetrative intercourse, and delayed detection of cervical or uterine pathologies when gynaecological exams are avoided due to pain.

Current management of PVD involves multidisciplinary teams (including physicians, psychologists, sex therapists, and physical therapists) aiming to change the vulvar pain experience through analgesia, cognitive reframing, PFM relaxation and/or stretching and the reduction of vulvar sensitivity. Multimodal physiotherapy (mPT), in the form of education, biofeedback, manual therapies, and the vaginal insertion of dilators is recommended in clinical guidelines as a first-line treatment for PVD. The investigators have published two studies on the effectiveness of mPT intervention for women with PVD; both with positive results; yet their impact was limited since they were preliminary - the first was a prospective cohort study and the second was a pilot randomized controlled trial (RCT). Elsewhere in the literature, the first large-scale RCT on mPT compared the effectiveness of mPT to topical lidocaine for pain reduction and improved sexual function among women with PVD. The results were very promising; 79% of females in a mPT group reported being much or very much improved compared with 39% in a topical lidocaine group, coincident with reporting reduced pain during intercourse and improved sexual function. However, due to the lack of a comparable control group, the evidence for mPT was rated as "low" in systematic reviews, highlighting the need for further research.

A different, and likely complementary, treatment avenue for PVD is to focus interventions on the vulvar tissues themselves. One therapeutic option is photobiomodulation (PBM, aka low-level laser therapy, cold laser). PBM involves irradiation of tissue with a combination of red and near infrared light. PBM is theorized to initiate a series of physiological reactions within the cells exposed to light at specific wavelengths, leading to the restoration of normal cell structure and function. Although the mechanisms of action of PBM are not fully understood, positive effects of PBM have been found in clinical populations with chronic neuropathic pain, including carpal tunnel syndrome and trigeminal neuralgia. Recent evidence shows elevated bradykinin signaling (one of the most potent inducers of inflammatory pain) on the surface of vestibular fibroblasts collected from sites of intense pain in patients with PVD. The fibroblasts, in turn, respond vigorously to bradykinin, producing IL-6, which has strong expression in numerous pain conditions. Given our current understanding of PVD pathophysiology, and the suspected mechanistic actions of PBM, this intervention may provide an effective, non-invasive, approach to the management of PVD through reducing inflammation, promoting cell repair, and producing anesthesia.

The available evidence suggests that both mPT and PBM may be effective interventions for PVD; it is plausible that combining these two therapies may result in an additive effect and may result in a more effective approach than either intervention alone. The investigators have just completed a sham-controlled pilot RCT (NCT04234542) using a comprehensive PBM intervention, and the results are extremely promising. Those who received the real PBM improved by 25% on the pain severity domain of the Vulvar Pain Assessment Questionnaire (VPAQ), which was significantly greater than the sham PBM group. They also reported significant improvements in emotional responses to pain and sexual interference relative to baseline. Thirty-eight percent of participants who received the real PBM intervention reported >30% improvement in their condition. And while the sham PBM group did not demonstrate significant reductions in pain sensitivity, the real PBM group demonstrated a 59% increase in pressure pain threshold (PPThresh) at the vulvar vestibule. A full RCT is clearly warranted.

The proposed trial will evaluate each intervention separately as well as a combined intervention group, as it is essential that we find effective, comprehensive, physiologically focused interventions that reduce vulvar pain severity and also improve the emotional, cognitive and functional burdens experienced by those who live with PVD. This will be a double-blind, multicenter RCT designed according to the Consolidated Standards of Reporting Trials (CONSORT) statement. The design will involve PBM (real, sham) and mPT (yes, no), resulting in four study groups: real PBM, sham PBM, PBM combined with mPT, and sham PBM combined with mPT. We did not include a sham mPT intervention due to existing RCT evidence supporting mPT's effectiveness, the lack of a validated sham mPT intervention for PVD, and the challenges in ensuring blinding with complex behavioral interventions like mPT.

mPT- The mPT protocol is largely based on the investigator's previously published protocol, including a greater focus on chronic pain education. It is very similar to that used in the RCT by Morin et al. (2021). At each site, the same physiotherapists (PTs) will provide all mPT treatments. The PTs have postgraduate certification in Women's Health physiotherapy, including advanced courses in pelvic pain, and >5 years of practice experience.

The goals of the mPT intervention are to educate the participant (vulvar anatomy and physiology, PVD pathophysiology, chronic pain pathophysiology, and self-care for chronic pain), increase flexibility of the tissue surrounding the vaginal opening, decrease pain sensitivity at the vulvar vestibule, decrease fear and anxiety towards vaginal penetration, increase control and relaxation of the PFMs upon vaginal penetration, and provide the participants with techniques to prevent and manage their vulvar pain. These goals are representative of clinical practice in Canada and the United States.

Participants will attend weekly mPT sessions for the first 8 weeks of the 14-week intervention period then every two weeks thereafter, for a total of 10 sessions. Sessions will last 45 minutes each, and, for combination therapy groups, will be scheduled wherever possible at the same visit as the PBM sessions described below. While standardized to a large extent, to approximate clinical practice, the protocol will be tailored to allow participants to progress at their own pace. For example, participants will only move up to the next dilator circumference when their pain on insertion is rated at ≤4/10 using the dilator they have been given. Participants will be offered the opportunity to bring a partner or other individual with them to a treatment session (8, 9 and/or 10) to learn how to perform basic manual stretches of the vagina that could be conducted before engaging in penetrative activities, and to receive further recommendations regarding pain and sexual activity. At the completion of the 14th treatment session, participants will be provided with a personalized home exercise program to continue on their own. At each mPT visit, adherence to the home program in the preceding week will be reported by the participant through an on-line portal (RedCAP) which is inaccessible to the PT to minimize reporting bias. Missed/cancelled mPT visits will be rescheduled wherever possible.

Real PBM/sham PBM- The PBM treatment protocol will be delivered through a Bioflex Laser Therapy (Toronto, Canada) system by the PT at each site. The participants and the PT delivering the PBM intervention will remain blinded to real/ sham PBM by having an independent researcher not involved in the study, program the real and the sham (all outputs set to 1%) PBM protocols into the PBM system, labelling one as protocol A the other as protocol B, while making program data inaccessible to the PT. This independent researcher will not disclose to participants or any member of the study team which protocol is real and which is sham until the end of the study, including following data analysis, with one exception. The study biostatistician will learn which group received the real vs sham PBM after completing the interim analysis only if the analysis reveals that the futility criteria may have been met; which will subsequently be disclosed to the Trial Steering Committee.

The precise PBM protocol, was developed in collaboration with the scientific advisor to BioFlex Laser Therapy and was used in the investigator's pilot RCT. Fifteen real/sham PBM treatments will be provided by the study PT over a 14- week period. The treatment is delivered in a progressive fashion, treating sites at the vulvar vestibule locally using a focal probe, and the perineum using an array. The dosage of the laser is increased progressively, while monitoring patient response and adjusting as necessary. Each treatment will last approximately 20 minutes and will be scheduled at the participant's convenience and in coordination with the mPT visits where relevant. Missed visits will be rescheduled wherever possible. Participants will progress through five treatment levels at their own rate. Patients randomized to the sham-PBM group will be offered the real PBM at the end of the study.

All groups - Regardless of assigned intervention group, participants will be asked not to engage in vaginal penetrative activities while undergoing the first 8 weeks of the intervention. After 8 weeks of the intervention period, participants will be advised that they may, if desired, engage in penetrative activities, both sexual and not (e.g., internal pelvic examination, tampon insertion), but to stop a given attempt if perceived pain exceeds a NRS of 4/10. This time point will coincide with an invitation being extended to the participant to invite a partner or other individual to participate in the mPT treatment. Adherence to all intervention visits (mPT, PBM) and any adverse events will be recorded by the study PT, the latter being reported to the NPA and the Trial Steering Committee within 2 days of occurrence.

Participants will be randomly allocated (1:1:1:1) to one of the four intervention groups using a concealed, computer-generated, permuted block randomization (block size= 4) stratified by PVD type (primary/ secondary) and site (Ottawa/ Quebec City) only after they have consented to participate and have completed the baseline assessment. The allocation sequence will be managed by an independent investigator not associated with the project. It will be concealed from the study team through storage in a password protected file on an encrypted computer, backed up in a password-protected directory on MSSharepoint. Group allocation will be revealed only to the recruitment officer, who will inform the PT who will deliver the intervention and the participant. Since all participants will be pre-menopausal, no stratification by age will be performed. While gender will be recorded and sub-analyses will be performed by gender if possible, the investigators will not stratify by gender because PVD prevalence by gender is unknown.

ELIGIBILITY:
Inclusion Criteria:

* Willing to travel to Ottawa area or Quebec City area
* Biologically born female older than eighteen years
* Pre-menopausal
* Not currently pregnant or pregnancy/given birth in the past six months
* Experiencing signs and symptoms consistent with provoked vestibulodynia alone or provoked vestibulodynia plus vaginismus

Exclusion Criteria:

* gynaecologist cannot insert a single digit intravaginally and thus the participant would be unlikely able to tolerate the assessment procedures
* other gynaecologic conditions such as lichen sclerosus, fissures, endometriosis, adenomyosis, or pelvic organ prolapse

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Vulvar Pain Assessment Questionnaire - Pain Severity | Baseline
  Developed by co-investigator Pukall and a subscale of the larger vulvar pain assessment questionnaire, participants report their average and worst vulvar pain intensity and associated unpleasantness and distress experienced during the previous four weeks. Scores are the the average of the items in the subscale, with the lowest possible score as 0 (Not at all) and the highest as 4 (very much). Higher score means worse symptoms
Vulvar Pain Assessment Questionnaire - Pain Severity | Within 2 weeks of the end of intervention
  Developed by co-investigator Pukall and a subscale of the larger vulvar pain assessment questionnaire, participants report their average and worst vulvar pain intensity and associated unpleasantness and distress experienced during the previous four weeks. Scores are the the average of the items in the subscale, with the lowest possible score as 0 (Not at all) and the highest as 4 (very much). Higher score means worse symptoms
Vulvar Pain Assessment Questionnaire - Pain Severity | 6 months post start of intervention
  Developed by co-investigator Pukall and a subscale of the larger vulvar pain assessment questionnaire, participants report their average and worst vulvar pain intensity and associated unpleasantness and distress experienced during the previous four weeks. Scores are the the average of the items in the subscale, with the lowest possible score as 0 (Not at all) and the highest as 4 (very much). Higher score means worse symptoms
Vulvar Pain Assessment Questionnaire - Pain Severity | 12 months post start of intervention
  Developed by co-investigator Pukall and a subscale of the larger vulvar pain assessment questionnaire, participants report their average and worst vulvar pain intensity and associated unpleasantness and distress experienced during the previous four weeks. Scores are the the average of the items in the subscale, with the lowest possible score as 0 (Not at all) and the highest as 4 (very much). Higher score means worse symptoms

SECONDARY OUTCOMES:
Tampon Test | Baseline
  A proxy measure of intercourse pain. This test involves the participant inserting and removing a non-lubricated regular Tampax tampon, then reporting their overall pain experience using a NRS (0=no pain; 10 = worst possible pain).
Tampon Test | Within 2 weeks of the end of the intervention
  A proxy measure of intercourse pain. This test involves the participant inserting and removing a non-lubricated regular Tampax tampon, then reporting their overall pain experience using a NRS (0=no pain; 10 = worst possible pain).
Tampon Test | 6 months post start of the intervention
  A proxy measure of intercourse pain. This test involves the participant inserting and removing a non-lubricated regular Tampax tampon, then reporting their overall pain experience using a NRS (0=no pain; 10 = worst possible pain).
Tampon Test | 12 months post start of the intervention
  A proxy measure of intercourse pain. This test involves the participant inserting and removing a non-lubricated regular Tampax tampon, then reporting their overall pain experience using a NRS (0=no pain; 10 = worst possible pain).
Provoked vulvar pain sensitivity | Baseline
  Vulvar pressure pain sensitivity will be measured using the investigators' custom electronic vulvalgesiometer (V-QueST), designed and validated specifically for quantitative sensory testing of the vulva. Force will be applied incrementally to the 3 o'clock, 6 o'clock and 9 o'clock position within the vulvar vestibule through a cotton swab interfaced with a force sensor, and the participant will be asked to indicate their pressure pain threshold (PPThresh) as well as the force at which the pain is no longer tolerable (PPTol). The median value across three trials will be retained as the outcome
Provoked vulvar pain sensitivity | 2 weeks post intervention
  Vulvar pressure pain sensitivity will be measured using the investigators' custom electronic vulvalgesiometer (V-QueST), designed and validated specifically for quantitative sensory testing of the vulva. Force will be applied incrementally to the 3 o'clock, 6 o'clock and 9 o'clock position within the vulvar vestibule through a cotton swab interfaced with a force sensor, and the participant will be asked to indicate their pressure pain threshold (PPThresh) as well as the force at which the pain is no longer tolerable (PPTol). The median value across three trials will be retained as the outcome
Provoked vulvar pain sensitivity | 6 months post start of the intervention
  Vulvar pressure pain sensitivity will be measured using the investigators' custom electronic vulvalgesiometer (V-QueST), designed and validated specifically for quantitative sensory testing of the vulva. Force will be applied incrementally to the 3 o'clock, 6 o'clock and 9 o'clock position within the vulvar vestibule through a cotton swab interfaced with a force sensor, and the participant will be asked to indicate their pressure pain threshold (PPThresh) as well as the force at which the pain is no longer tolerable (PPTol). The median value across three trials will be retained as the outcome
Provoked vulvar pain sensitivity | 12 months post start of the intervention
  Vulvar pressure pain sensitivity will be measured using the investigators' custom electronic vulvalgesiometer (V-QueST), designed and validated specifically for quantitative sensory testing of the vulva. Force will be applied incrementally to the 3 o'clock, 6 o'clock and 9 o'clock position within the vulvar vestibule through a cotton swab interfaced with a force sensor, and the participant will be asked to indicate their pressure pain threshold (PPThresh) as well as the force at which the pain is no longer tolerable (PPTol). The median value across three trials will be retained as the outcome
Vulvar pain assessment questionnaire - full inventory | Baseline
  The other subscales of the VPAQ are designed to assess emotional response, cognitive response, life interference, sexual function interference and self-stimulation/penetration interference associated with vulvar pain, which are all recommended to capture different aspects of the pain experience among those with PVD. Each subscale is scored separately and is the average of the items. The lowest possible score is 0 (Not at all) and the highest is 4 (very much). Higher score means worse symptoms.
Vulvar pain assessment questionnaire - full inventory | Within 2 weeks post intervention
  The other subscales of the VPAQ are designed to assess emotional response, cognitive response, life interference, sexual function interference and self-stimulation/penetration interference associated with vulvar pain, which are all recommended to capture different aspects of the pain experience among those with PVD. Each subscale is scored separately and is the average of the items. The lowest possible score is 0 (Not at all) and the highest is 4 (very much). Higher score means worse symptoms.
Vulvar pain assessment questionnaire - full inventory | 6 months post start of the intervention
  The other subscales of the VPAQ are designed to assess emotional response, cognitive response, life interference, sexual function interference and self-stimulation/penetration interference associated with vulvar pain, which are all recommended to capture different aspects of the pain experience among those with PVD. Each subscale is scored separately and is the average of the items. The lowest possible score is 0 (Not at all) and the highest is 4 (very much). Higher score means worse symptoms.
Vulvar pain assessment questionnaire - full inventory | 12 months post start of the intervention
  The other subscales of the VPAQ are designed to assess emotional response, cognitive response, life interference, sexual function interference and self-stimulation/penetration interference associated with vulvar pain, which are all recommended to capture different aspects of the pain experience among those with PVD. Each subscale is scored separately and is the average of the items. The lowest possible score is 0 (Not at all) and the highest is 4 (very much). Higher score means worse symptoms.
Pain Catastrophizing Scale | Baseline
  A reliable and valid scale to measure of catastrophizing of pain. The scores from this questionnaire is predictors of intensity of physical and emotional distress. It is a self-report measure, consisting of 13 items scored from 0 to 4, resulting in a total possible score of 52. The higher the score, the more catastrophizing thoughts are present.
Pain Catastrophizing Scale | Within 2 weeks post-intervention
  A reliable and valid scale to measure of catastrophizing of pain. The scores from this questionnaire is predictors of intensity of physical and emotional distress. It is a self-report measure, consisting of 13 items scored from 0 to 4, resulting in a total possible score of 52. The higher the score, the more catastrophizing thoughts are present.
Pain Catastrophizing Scale | 6 months post start of intervention
  A reliable and valid scale to measure of catastrophizing of pain. The scores from this questionnaire is predictors of intensity of physical and emotional distress. It is a self-report measure, consisting of 13 items scored from 0 to 4, resulting in a total possible score of 52. The higher the score, the more catastrophizing thoughts are present.
Pain Catastrophizing Scale | 12-months post start of intervention
  A reliable and valid scale to measure of catastrophizing of pain. The scores from this questionnaire is predictors of intensity of physical and emotional distress. It is a self-report measure, consisting of 13 items scored from 0 to 4, resulting in a total possible score of 52. The higher the score, the more catastrophizing thoughts are present.
Female sexual function index | Baseline
  This is a 19-item validated questionnaire for assessing the key dimension of sexual function in women, considered a gold standard for evaluation of sexual function. It assesses six domains: desire, arousal , lubrification, orgasm, satisfaction, and pain. All scores are totaled for a maximum of 36. Higher scores represents better sexual function. A score ≤26.55 has been set as a cutoff to identify those at risk for sexual dysfunction.
Female sexual function index | Within 2 weeks post intervention
  This is a 19-item validated questionnaire for assessing the key dimension of sexual function in women, considered a gold standard for evaluation of sexual function. It assesses six domains: desire, arousal , lubrification, orgasm, satisfaction, and pain. All scores are totaled for a maximum of 36. Higher scores represents better sexual function. A score ≤26.55 has been set as a cutoff to identify those at risk for sexual dysfunction.
Female sexual function index | 6 months post start of intervention
  This is a 19-item validated questionnaire for assessing the key dimension of sexual function in women, considered a gold standard for evaluation of sexual function. It assesses six domains: desire, arousal , lubrification, orgasm, satisfaction, and pain. All scores are totaled for a maximum of 36. Higher scores represents better sexual function. A score ≤26.55 has been set as a cutoff to identify those at risk for sexual dysfunction.
Female sexual function index | 12 months post start of intervention
  This is a 19-item validated questionnaire for assessing the key dimension of sexual function in women, considered a gold standard for evaluation of sexual function. It assesses six domains: desire, arousal , lubrification, orgasm, satisfaction, and pain. All scores are totaled for a maximum of 36. Higher scores represents better sexual function. A score ≤26.55 has been set as a cutoff to identify those at risk for sexual dysfunction.
Central sensitization inventory | Baseline
  A self-reported outcome measure designed to identify patients who have symptoms that may be related to central sensitisation (CS) or central sensitivity syndromes (CSS). Part A includes 25 questions related to common CSS symptoms.
  Part B determines if the patient has been diagnosed with certain CSS disorders or related disorders, such as anxiety and depression. CSI severity levels have been established for part A: subclinical = 0 to 29; mild = 30 to 39; moderate = 40 to 49; severe = 50 to 59; and extreme = 60 to 100.
Central sensitization inventory | Within 2 weeks post-intervention
  A self-reported outcome measure designed to identify patients who have symptoms that may be related to central sensitisation (CS) or central sensitivity syndromes (CSS). Part A includes 25 questions related to common CSS symptoms.
  Part B determines if the patient has been diagnosed with certain CSS disorders or related disorders, such as anxiety and depression. CSI severity levels have been established for part A: subclinical = 0 to 29; mild = 30 to 39; moderate = 40 to 49; severe = 50 to 59; and extreme = 60 to 100.
Central sensitization inventory | 6 months post start of intervention,
  A self-reported outcome measure designed to identify patients who have symptoms that may be related to central sensitisation (CS) or central sensitivity syndromes (CSS). Part A includes 25 questions related to common CSS symptoms.
  Part B determines if the patient has been diagnosed with certain CSS disorders or related disorders, such as anxiety and depression. CSI severity levels have been established for part A: subclinical = 0 to 29; mild = 30 to 39; moderate = 40 to 49; severe = 50 to 59; and extreme = 60 to 100.
Central sensitization inventory | 12 months post start of intervention
  A self-reported outcome measure designed to identify patients who have symptoms that may be related to central sensitisation (CS) or central sensitivity syndromes (CSS). Part A includes 25 questions related to common CSS symptoms.
  Part B determines if the patient has been diagnosed with certain CSS disorders or related disorders, such as anxiety and depression. CSI severity levels have been established for part A: subclinical = 0 to 29; mild = 30 to 39; moderate = 40 to 49; severe = 50 to 59; and extreme = 60 to 100.
Chronic Pain Acceptance Questionnaire | Baseline
  A self-report measure designed to assess the degree to which individuals with chronic pain accept their pain and engage in life activities despite it. It evaluates two key components: pain willingness (the ability to experience pain without trying to control or avoid it) and activity engagement (the extent to which a person participates in life activities regardless of pain). The CPAQ uses a 7-point Likert scale ranging from 0 (never true) to 6 (always true), with higher scores suggesting a greater level of acceptance of chronic pain.
Chronic Pain Acceptance Questionnaire | 2 weeks post intervention
  A self-report measure designed to assess the degree to which individuals with chronic pain accept their pain and engage in life activities despite it. It evaluates two key components: pain willingness (the ability to experience pain without trying to control or avoid it) and activity engagement (the extent to which a person participates in life activities regardless of pain). The CPAQ uses a 7-point Likert scale ranging from 0 (never true) to 6 (always true), with higher scores suggesting a greater level of acceptance of chronic pain.
Chronic Pain Acceptance Questionnaire | 6 months post start of the intervention
  A self-report measure designed to assess the degree to which individuals with chronic pain accept their pain and engage in life activities despite it. It evaluates two key components: pain willingness (the ability to experience pain without trying to control or avoid it) and activity engagement (the extent to which a person participates in life activities regardless of pain). The CPAQ uses a 7-point Likert scale ranging from 0 (never true) to 6 (always true), with higher scores suggesting a greater level of acceptance of chronic pain.
Chronic Pain Acceptance Questionnaire | 12 months post start of the intervention
  A self-report measure designed to assess the degree to which individuals with chronic pain accept their pain and engage in life activities despite it. It evaluates two key components: pain willingness (the ability to experience pain without trying to control or avoid it) and activity engagement (the extent to which a person participates in life activities regardless of pain). The CPAQ uses a 7-point Likert scale ranging from 0 (never true) to 6 (always true), with higher scores suggesting a greater level of acceptance of chronic pain.
Non-sexual insertional pain | Baseline
  A single self-reported question through which participants provide a ordinal rating from 0 (no pain) to 10 (maximum pain) based on their perceived pain during non-sexual vaginal insertion.
Non-sexual insertional pain | 2 weeks post intervention
  A single self-reported question through which participants provide a ordinal rating from 0 (no pain) to 10 (maximum pain) based on their perceived pain during non-sexual vaginal insertion.
Non-sexual insertional pain | 6 months post start of the intervention
  A single self-reported question through which participants provide a ordinal rating from 0 (no pain) to 10 (maximum pain) based on their perceived pain during non-sexual vaginal insertion.
Non-sexual insertional pain | 12 months post start of the intervention
  A single self-reported question through which participants provide a ordinal rating from 0 (no pain) to 10 (maximum pain) based on their perceived pain during non-sexual vaginal insertion.
Sexual Insertion pain | Baseline
  A single self-reported question through which participants provide a ordinal rating from 0 (no pain) to 10 (maximum pain) based on their perceived pain during sexual vaginal penetration.
Sexual Insertion pain | 2 weeks post intervention
  A single self-reported question through which participants provide a ordinal rating from 0 (no pain) to 10 (maximum pain) based on their perceived pain during sexual vaginal penetration.
Sexual Insertion pain | 6 months post start of the intervention
  A single self-reported question through which participants provide a ordinal rating from 0 (no pain) to 10 (maximum pain) based on their perceived pain during sexual vaginal penetration.
Sexual Insertion pain | 12 months post start of the intervention
  A single self-reported question through which participants provide a ordinal rating from 0 (no pain) to 10 (maximum pain) based on their perceived pain during sexual vaginal penetration.
Patient global impression of change | 2 weeks post intervention
  A self-reported measure about patients' belief on treatment efficacy. The PGIC is a 7 point likert scale rating improvement from "very much worse" (7) to "very much improved" (1).
Patient global impression of change | 6 months post start of intervention
  A self-reported measure about patients' belief on treatment efficacy. The PGIC is a 7 point likert scale rating improvement from "very much worse" (7) to "very much improved" (1).
Patient global impression of change | 12 months post start of intervention
  A self-reported measure about patients' belief on treatment efficacy. The PGIC is a 7 point likert scale rating improvement from "very much worse" (7) to "very much improved" (1).

CONTACTS AND LOCATIONS:
Overall Officials: Linda McLean, PhD, Principal Investigator — University of Ottawa; Stephanie Bernard, PhD, Principal Investigator — University of Laval
Locations (2):
- Canada (2):
  - Motor Function Measurement Lab, Ottawa, Ontario
  - Bernard Lab, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Participant data will be anonymized using ID numbers and stored on spreadsheets. Spreadsheets will be provided by email upon request and based on the planned use of the data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available for 10 years after the publication of the study results.
Access Criteria: Planned use of data for systematic review or meta-analysis.

REFERENCES:
- [Background] Dargie E, Holden RR, Pukall CF. The Vulvar Pain Assessment Questionnaire: Factor Structure, Preliminary Norms, Internal Consistency, and Test-Retest Reliability. J Sex Med. 2017 Dec;14(12):1585-1596. doi: 10.1016/j.jsxm.2017.10.072. PMID 29198513
- [Background] Vowles KE, Kruger ES, Bailey RW, Sowden G, Ashworth J, Hickman J, McCracken LM. Initial evaluation of the Chronic Pain Acceptance Questionnaire - 2. Eur J Pain. 2020 Nov;24(10):2027-2036. doi: 10.1002/ejp.1650. Epub 2020 Sep 21. PMID 32816389
- [Background] Vandyken C, Hilton S. Physical Therapy in the Treatment of Central Pain Mechanisms for Female Sexual Pain. Sex Med Rev. 2017 Jan;5(1):20-30. doi: 10.1016/j.sxmr.2016.06.004. Epub 2016 Aug 3. PMID 27498209
- [Background] LePage K, Selk A. What Do Patients Want? A Needs Assessment of Vulvodynia Patients Attending a Vulvar Diseases Clinic. Sex Med. 2016 Dec;4(4):e242-e248. doi: 10.1016/j.esxm.2016.06.003. Epub 2016 Jul 30. PMID 27484917
- [Background] Bergeron S, Binik YM, Khalife S, Pagidas K, Glazer HI, Meana M, Amsel R. A randomized comparison of group cognitive--behavioral therapy, surface electromyographic biofeedback, and vestibulectomy in the treatment of dyspareunia resulting from vulvar vestibulitis. Pain. 2001 Apr;91(3):297-306. doi: 10.1016/S0304-3959(00)00449-8. PMID 11275387
- [Background] Lev-Sagie A, Kopitman A, Brzezinski A. Low-Level Laser Therapy for the Treatment of Provoked Vestibulodynia-A Randomized, Placebo-Controlled Pilot Trial. J Sex Med. 2017 Nov;14(11):1403-1411. doi: 10.1016/j.jsxm.2017.09.004. Epub 2017 Sep 29. PMID 28970071
- [Background] Dargie EE, Chamberlain SM, Pukall CF. Provoked Vestibulodynia: Diagnosis, Self-Reported Pain, and Presentation During Gynaecological Examinations. J Obstet Gynaecol Can. 2017 Mar;39(3):145-151. doi: 10.1016/j.jogc.2017.01.001. PMID 28343555
- [Background] McLean L, Thibault-Gagnon S, Brooks K, Goldfinger C, Pukall C, Chamberlain S. Differences in Pelvic Morphology Between Women With and Without Provoked Vestibulodynia. J Sex Med. 2016 Jun;13(6):963-71. doi: 10.1016/j.jsxm.2016.04.066. PMID 27215690
- [Background] Morin M, Bergeron S, Khalife S, Mayrand MH, Binik YM. Morphometry of the pelvic floor muscles in women with and without provoked vestibulodynia using 4D ultrasound. J Sex Med. 2014 Mar;11(3):776-85. doi: 10.1111/jsm.12367. Epub 2013 Nov 6. PMID 24344835
- [Background] Gentilcore-Saulnier E, McLean L, Goldfinger C, Pukall CF, Chamberlain S. Pelvic floor muscle assessment outcomes in women with and without provoked vestibulodynia and the impact of a physical therapy program. J Sex Med. 2010 Feb;7(2 Pt 2):1003-22. doi: 10.1111/j.1743-6109.2009.01642.x. Epub 2010 Jan 6. PMID 20059663
- [Background] Reissing ED, Brown C, Lord MJ, Binik YM, Khalife S. Pelvic floor muscle functioning in women with vulvar vestibulitis syndrome. J Psychosom Obstet Gynaecol. 2005 Jun;26(2):107-13. doi: 10.1080/01443610400023106. PMID 16050536
- [Background] Mayer TG, Neblett R, Cohen H, Howard KJ, Choi YH, Williams MJ, Perez Y, Gatchel RJ. The development and psychometric validation of the central sensitization inventory. Pain Pract. 2012 Apr;12(4):276-85. doi: 10.1111/j.1533-2500.2011.00493.x. Epub 2011 Sep 27. PMID 21951710
- [Background] Meyer-Bahlburg HF, Dolezal C. The female sexual function index: a methodological critique and suggestions for improvement. J Sex Marital Ther. 2007 May-Jun;33(3):217-24. doi: 10.1080/00926230701267852. PMID 17454519
- [Background] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Background] Pukall CF, Young RA, Roberts MJ, Sutton KS, Smith KB. The vulvalgesiometer as a device to measure genital pressure-pain threshold. Physiol Meas. 2007 Dec;28(12):1543-50. doi: 10.1088/0967-3334/28/12/008. Epub 2007 Dec 3. PMID 18057518
- [Background] Goldstein AT, Pukall CF, Brown C, Bergeron S, Stein A, Kellogg-Spadt S. Vulvodynia: Assessment and Treatment. J Sex Med. 2016 Apr;13(4):572-90. doi: 10.1016/j.jsxm.2016.01.020. Epub 2016 Mar 25. PMID 27045258
- [Background] Spoelstra SK, Dijkstra JR, van Driel MF, Weijmar Schultz WC. Long-term results of an individualized, multifaceted, and multidisciplinary therapeutic approach to provoked vestibulodynia. J Sex Med. 2011 Feb;8(2):489-96. doi: 10.1111/j.1743-6109.2010.01941.x. PMID 20646179
- [Background] Harlow BL, Stewart EG. A population-based assessment of chronic unexplained vulvar pain: have we underestimated the prevalence of vulvodynia? J Am Med Womens Assoc (1972). 2003 Spring;58(2):82-8. PMID 12744420